CLINICAL TRIAL: NCT05393726
Title: Ultrasound-Guided Suprainguinal Fascia Iliaca Block Versus Lumbar Erector Spinae Plane Block for Oncologic Thigh Surgery: A Randomized Controlled Trial
Brief Title: Suprainguinal Fascia Iliaca Block Versus Lumbar Erector Spinae Plane Block for Oncologic Thigh Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Hamed Sayed Ashour, assistant lecturer, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2203-301-014
Record Dates: First submitted 2022-05-22; First posted 2022-05-26 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Perioperative Pain
Keywords: Suprainguinal Fascia Iliaca Block; Lumbar Erector Spinae Plane Block; postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Suprainguinal Fascia Iliaca Block group (Experimental): Patients will receive ultrasound-guided suprainguinal fascia iliaca block injection 40 ml of bupivacaine 0.25% mixed with 2 ml of dexamethasone 4 mg/ml.
  Interventions: Procedure: Ultrasound-Guided Suprainguinal Fascia Iliaca Block Versus Lumbar Erector Spinae Plane Block
- Lumbar Erector Spinae Plane Block group (Experimental): Patients will receive ultrasound-guided lumber erector spinae plane block (L-ESPB) injection 40ml bupivacaine 0.25% mixed with 2 ml of dexamethasone 4 mg/ml.
  Interventions: Procedure: Ultrasound-Guided Suprainguinal Fascia Iliaca Block Versus Lumbar Erector Spinae Plane Block
- control group (No Intervention): Patients underwent surgery under general anesthesia and received the perioperative routine protocol of analgesia by using I.V. fentanyl (1µg/kg), with elevation of mean arterial blood pressure for more than 20% of their baseline values, additional bolus doses of fentanyl 0.5 µg /kg.

INTERVENTIONS:
Procedure: Ultrasound-Guided Suprainguinal Fascia Iliaca Block Versus Lumbar Erector Spinae Plane Block — Suprainguinal Fascia Iliaca Block group will receive ultrasound-guided suprainguinal fascia iliaca block injection 40 ml of bupivacaine 0.25% mixed with 2 ml of dexamethasone 4 mg/ml.
  Lumbar Erector Spinae Plane Block group will receive ultrasound-guided lumber erector spinae plane block (L-ESPB) injection 40 ml bupivacaine 0.25% mixed with 2 ml of dexamethasone 4 mg/ml.
  control group will underwent surgery under general anesthesia and receive the perioperative routine protocol of analgesia
  Arms: Lumbar Erector Spinae Plane Block group; Suprainguinal Fascia Iliaca Block group

SUMMARY:
This is a prospective; double blinded randomized controlled trial that will be conducted on cancer patients subjected to oncologic thigh surgery.The aim of this study is to evaluate and compare the analgesic effect of supra-inguinal fascia iliaca block and lumbar erector spinae plane block in oncologic thigh surgery.Patients will be randomized into three equal comparable groups, Group A (Ultrasound-guided supra-inguinal fascia iliaca block (SIFIB)), Group B (Ultrasound-guided lumbar erector spinae plane block (L-ESPB)), and Group C (control group). Primary outcome parameter is the total postoperative morphine consumption over the first 24 hours postoperative. Data will be analyzed using IBM SPSS 26 (SPSS Inc., Chicago, IL).

DETAILED DESCRIPTION:
Pain is one of the most common and significant postoperative events experienced by many surgical patients. Orthopedic surgery is a relatively painful surgery due to the significant amount of bone and soft tissue resection, damage, and reconstruction. After thigh surgery for sarcomas, the patient may experience any of three distinct types of pain, including acute postoperative pain, persistent long-term nociceptive pain, and neuropathic pain related to intraoperative nerve injuries. The management of pain in limb sparing surgery patients and amputated patients is crucial during the rehabilitation program and often its approach is multidisciplinary. The ultrasound-guided supra-inguinal fascia iliaca block further built on earlier anatomic discoveries to more reliably anesthetize the three nerves: femoral, lateral femoral cutaneous, and obturator. The supra-inguinal fascia iliaca block has evolved as an effective means of providing analgesia to the thigh, the knee, and, most notably, the hip. Ultrasound-guided erector spinae plane block (ESPB) is an interfascial plane block reported in the treatment of postoperative pain from surgical procedures, ranging from shoulder to hip surgery. When performed at the lumbar 4th vertebral level, ESPB led to sensorial blockage between Th12 and L4 dermatomes lead to effective postoperative analgesia in hip and proximal femoral surgery. Although supra-inguinal fascia iliaca block and L-ESPB successfully reduced postoperative opioid consumption in previous study, no study has ever compared their efficacy in postoperative analgesia of adult patients undergoing oncologic thigh surgery under general anesthesia. Thus, in this randomized comparative study we are aiming to fill this gape in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65 years.
* Physical status: ASA II,III
* Patient undergoing oncologic thigh surgery under general anesthesia.
* Body mass index (BMI): 20-40 kg/m 2

Exclusion Criteria:

* Patient refusal.
* Sensitivity or contraindication to local anesthetics.
* Bleeding tendency due to coagulopathy.
* Patients with opioid dependence or alcohol or drug abuse.
* Patients with psychiatric illness that prevent them from proper perception and assessment of pain.
* Contraindication to regional anesthesia e.g. local infection at the site of block, coagulopathy with INR more than 1.6: hereditary (e.g. hemophilia, fibrinogen abnormalities & deficiency factor II) acquired (e.g. impaired liver functions with PC less than 60%, vitamin K deficiency & therapeutic anticoagulant drugs) .
* Significant renal insufficiency (plasma creatinine more than 1.5 mg/dl).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
postoperative morphine consumption . | over the first 24 hours postoperative
  Total postoperative morphine consumption over the first 24 hours postoperative.

SECONDARY OUTCOMES:
fentanyl consumption. | intra-operative
  Total intra-operative fentanyl consumption.
The time of first rescue analgesia. | over the first 24 hours postoperative
  The time of first rescue analgesia.
Visual Analogue Scale | over the first 24 hours postoperative
  Pain will be assessed using Visual Analogue Scale, both at rest and during movement, pain scores using visual Analogue Scale will be recorded in the post anesthesia care unit and for the next 24 hours postoperative.score (0) means no pain, scores(1-3) are considered mild pain, (4-6) moderate pain and (7-10) severe pain

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt